CLINICAL TRIAL: NCT00534131
Title: A Multicentre Trial of the Anterior Perineal PlanE for Ultra Low Anterior Resection of the Rectum (The APPEAR Technique) in the Prevention of Permanent Stoma in Benign and Malignant Disease
Brief Title: Anterior Perineal Plane for Ultra Low Anterior Resection of the Rectum
Acronym: APPEAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09/H0704/30
Record Dates: First submitted 2007-09-21; First posted 2007-09-24 (Estimated); Last update posted 2023-03-01 (Actual); Status verified 2008-06

CONDITIONS: Rectal Neoplasms; Colitis, Ischemic; Colitis, Ulcerative
MeSH Terms: conditions — Rectal Neoplasms; Colitis, Ischemic; Colitis, Ulcerative | interventions — Proctectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm 1 (Active Comparator): Patients for whom a standard abdominal approach is adequate to excise the distal third of the rectum (without jeopardising oncological clearance if appropriate).
  Interventions: Procedure: Standard abdominal approach for rectal excision
- Arm 2 (Experimental): Combined abdominal and trans-perineal approach to excise the distal third of the rectum, while preserving the anal canal
  Interventions: Procedure: APPEAR Procedure
- Arm 3 (Active Comparator): Standard proctectomy to excise the distal third of the rectum and the anal canal
  Interventions: Procedure: Proctectomy

INTERVENTIONS:
Procedure: Standard abdominal approach for rectal excision — Standard abdominal approach for rectal excision
  Arms: Arm 1
Procedure: APPEAR Procedure — Perineal incision to reach the distal rectum
  Other Names: Anterior Perineal PlanE for ultra low rectal excision
  Arms: Arm 2
Procedure: Proctectomy — standard rectal excision which does not preserve the anal canal
  Arms: Arm 3

SUMMARY:
Anal sphincter preserving operations are now commonplace for both cancer and non-cancerous rectal diseases. However, this has not always been the case and this development has been facilitated by the invention of circular stapling instruments, which allow the bowel to be reconnected to the anal sphincters, where it would almost be impossible to do so manually. Nevertheless, some patients still require a permanent ostomy, as even with stapling devices ultra low joins of the bowel and sphincter muscles cannot always be performed by a conventional surgery. Therefore, a variety of alternative techniques have been proposed to avoid a permanent ostomy, but these have not become widespread due to the technical difficulty in performing them, their failure to completely eradicate rectal disease, and the damage they inflict upon the anal sphincters resulting in poor bowel function after surgery.

The ideal ultra low sphincter preserving operation should remove the rectal disease entirely, allow the small or large bowel to be safely joined to the anal sphincters under direct vision, and retain the sphincter mechanism in its entirety. We propose such a technique that we term the APPEAR procedure, which approaches the lower third of the rectum via an incision between the scrotum or vagina, and the anal sphincters. This procedure preserves sphincter integrity, and allows either a stapled or manual join of the bowel to the sphincter mechanism, under direct vision. This trial is being conducted as a pilot study, with the procedure only offered to patients for whom a conventional sphincter saving procedure was technically impossible, or contraindicated.

DETAILED DESCRIPTION:
This study is recruiting patients with distal third rectal pathology, for whom a conventional sphincter saving procedure is contraindicated, or likely to be technically impossible.

Recruited patients will initially undergo trial dissection by conventional sphincter preserving surgical techniques, which if successful will result in patients entering study arm 1.

However, should this not be possible, a trial anterior perineal dissection will be attempted, with patients entered into study arm 2 if perineal dissection is adequate to allow full rectal excision, and preserve sphincter integrity.

If during a trial of anterior perineal dissection it is decided that sphincter preservation is not safe, or will not allow eradication of rectal disease, conventional proctectomy will be performed, with patients entering study arm 3.

ELIGIBILITY:
Inclusion Criteria:

* All patients regardless of sex
* Undergoing surgery (with curative intent) to excise the lower third of the rectum who may require a permanent stoma
* Deemed suitable by multidisciplinary team.

Exclusion Criteria:

* Patients under the age of 16
* Patients in whom sphincter preservation has already been deemed inappropriate for medical or surgical reasons (e.g. by an MDT for oncological cure), or in whom surgery has been deemed generally inappropriate.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-04-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-11-01 (Actual)

PRIMARY OUTCOMES:
Yield (within each arm of study) | 5 years
Functional assessment (faecal continence) | 5 years
Surgical Safety Assessment | 1 year
Oncological safety assessment - where appropriate | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Prof Norman S Williams, MS FRCS, Study Chair — Centre for Academic Surgery, Queen Mary University of London; Charles H Knowles, PhD FRCS, Study Director — Centre for Academic Surgery, Queen Mary University of London; Khalid El-Gendy, MBBS MRCS, Principal Investigator — Centre for Academic Surgery, Queen Mary University of London
Locations (1):
- Centre For Academic Surgery, The Royal London Hospital, London, England, United Kingdom

REFERENCES:
- [Derived] Williams NS, Murphy J, Knowles CH. Anterior Perineal PlanE for Ultra-low Anterior Resection of the Rectum (the APPEAR technique): a prospective clinical trial of a new procedure. Ann Surg. 2008 May;247(5):750-8. doi: 10.1097/SLA.0b013e31816b2ee3. PMID 18438111